CLINICAL TRIAL: NCT04764851
Title: A Phase 1, Open-Label, Fixed Sequence Drug-Drug Interaction Study to Evaluate the Effects of Repeat Doses of Ecopipam on the Pharmacokinetics of Multiple Substrates for Drug Metabolism and Transport in Healthy Subjects
Brief Title: Drug-Drug Interaction Study to Evaluate the Effects of Ecopipam on the Pharmacokinetics of Multiple Substrates
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: A number of subjects withdrew consent leaving the study without adequate power to achieve its primary end points.
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Syneos Health (Other); Nuventra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EBS-101-HV-101
Record Dates: First submitted 2021-01-18; First posted 2021-02-21 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Drug-Interactions

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Other): ecopipam HCl oral tablets of 12.5, 50, 75, and 100 mg daily for up to 20 days
  Cohort 1 Probe Cocktail given on 2 separate days:
  * midazolam: 1 µg infused IV
  * caffeine: 200 mg oral tablet
  * omeprazole: two 20 mg oral tablets
  * dextromethorphan: 1.6mL (containing ~10 mg) oral solution
  Interventions: Drug: ecopipam HCl ~2mg/kg/day; Combination Product: Cohort 1 Probe Cocktail
- Cohort 2 (Other): ecopipam HCl oral tablets of 12.5, 50, 75, and 100 mg daily for up to 20 days
  Cohort 2 Probe Cocktail given on 3 separate days:
  * midazolam: 10 µg/mL given as 1mL oral solution.
  * dabigatran: 375 µg/mL and pitavastatin: 10 µg/mL given as 1mL oral solution
  * rosuvastatin: 25 µg/mL and atorvastatin: 50 µg/mL given as 2mL oral solution
  Interventions: Drug: ecopipam HCl ~2mg/kg/day; Combination Product: Cohort 2 Probe Cocktail
- Cohort 3 (Other): ecopipam HCl oral tablets of 12.5, 50, 75, and 100 mg daily for up to 20 days
  Cohort 3 Probe Cocktail given on 2 separate days:
  - bupropion: 100mg oral tablet
  Interventions: Drug: ecopipam HCl ~2mg/kg/day; Combination Product: Cohort 3 Probe Cocktail

INTERVENTIONS:
Drug: ecopipam HCl ~2mg/kg/day — oral tablet
Combination Product: Cohort 1 Probe Cocktail — dextromethorphan, caffeine, omeprazole, and midazolam
  Arms: Cohort 1
Combination Product: Cohort 2 Probe Cocktail — dabigatran, pitavastatin, rosuvastatin, atorvastatin, midazolam
  Arms: Cohort 2
Combination Product: Cohort 3 Probe Cocktail — bupropion
  Arms: Cohort 3

SUMMARY:
This is a single center, open-label, fixed sequence Phase 1, drug-drug interaction (DDI) study in healthy subjects.

DETAILED DESCRIPTION:
Following a screening period of up to 28 days, subjects will be admitted to the clinical research unit into one of three cohorts. On the morning of Day 1, subjects in cohorts 1, 2, and 3 will receive fasted doses of probe substrate(s) per assigned cohort. On Day 5, Cohort 2 only will receive a second fasted dose of probe substrates. Subjects in cohorts 1, 2, and 3 will receive the final fasted dose of probe substrate(s) on Day 13. Fasted ecopipam administration will begin on Day 5 and will continue through Day 17 at ~2mg/kg for all cohorts. Ecopipam doses will be tapered starting on Day 18 by 25 mg/day increments until subjects are off drug, with final discharge occurring 24 hours after the ecopipam HCl dose has been reduced to 25 mg (Day 21, 23, or 25).

ELIGIBILITY:
Inclusion Criteria:

* Male subjects or female subjects of non-childbearing potential
* ≥18 and <55 years of age at the time of consent
* BMI >18.5 and <30 kg/m2 and a weight of ≥50 kg for males or ≥45 kg for females
* Sexually active males must use a double barrier method of contraception during the study and for at least 90 days after the last dose of study drug
* Male subjects must be willing not to donate sperm until 90 days following the last study drug administration

Exclusion Criteria:

* Personal or family History of significant medical illness
* Clinically significant abnormalities on screening tests/exams
* History of or significant risk of committing suicide
* Donation of plasma within 7 days prior to dosing
* Donation or significant loss of blood within 30 days prior to the first dosing
* Major surgery within 3 months or minor surgery within 1 month prior to admission
* Use of prohibited prescription, over-the-counter medications or natural health products
* Alcohol-based products 24 hours prior to admission
* Female subjects who are currently pregnant or lactating
* Positive pregnancy test
* Use of tobacco or nicotine products within 3 months prior to Screening
* Significant alcohol consumption
* History of drug abuse within the previous 2 years, or a positive drug screen
* History of allergy to study medications
* Undergoing abrupt discontinuation of alcohol or sedatives
* Not suitable for study in the opinion of the Principal Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Cmax of dextromethorphan (and its dextrorphan metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of dextromethorphan (and its dextrorphan metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax oral midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of dabigatran in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of dabigatran in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of pitavastatin (and its pitavastatin lactone metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of pitavastatin (and its pitavastatin lactone metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of rosuvastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of rosuvastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of dextromethorphan (and its dextrorphan metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of dextromethorphan (and its dextrorphan metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of dabigatran in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of dabigatran in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of pitavastatin (and its pitavastatin lactone metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of pitavastatin (and its pitavastatin lactone metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUCinf of rosuvastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUCinf of rosuvastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUCinf of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUCinf of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of dextromethorphan (and its dextrorphan metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of dextromethorphan (and its dextrorphan metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of IV midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of oral midazolam (and its 1'-hydroxymidazolam metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of dabigatran in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of dabigatran in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of pitavastatin (and its pitavastatin lactone metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of pitavastatin (and its pitavastatin lactone metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of rosuvastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of rosuvastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic
AUClast of atorvastatin (and its 4'-hydroxy atorvastatin metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic

SECONDARY OUTCOMES:
Cmax of bupropion (and its 4-hydroxybupropion metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of bupropion (and its 4-hydroxybupropion metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of caffeine (and its metabolite paraxanthine) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of caffeine (and its metabolite paraxanthine) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax omeprazole (and its 5'-hydroxy omeprazole metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax omeprazole (and its 5'-hydroxy omeprazole metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of bupropion (and its 4-hydroxybupropion metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of bupropion (and its 4-hydroxybupropion metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of caffeine (and its metabolite paraxanthine) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of caffeine (and its metabolite paraxanthine) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUCinf of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of bupropion (and its 4-hydroxybupropion metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of bupropion (and its 4-hydroxybupropion metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of caffeine (and its metabolite paraxanthine) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of caffeine (and its metabolite paraxanthine) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
AUClast of omeprazole (and its 5'-hydroxy omeprazole metabolite) in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dextromethorphan in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dextromethorphan in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for IV midazolam in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for IV midazolam in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for oral midazolam in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for oral midazolam in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dabigatran in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for dabigatran in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for pitavastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for pitavastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for rosuvastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for rosuvastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for atorvastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for atorvastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for bupropion in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for bupropion in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for caffeine in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for caffeine in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for omeprazole in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
CL/F for omeprazole in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dextromethorphan in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dextromethorphan in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for IV midazolam in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for IV midazolam in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for oral midazolam in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for oral midazolam in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dabigatran in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for dabigatran in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for pitavastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for pitavastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for rosuvastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for rosuvastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for atorvastatin in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for atorvastatin in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for bupropion in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for bupropion in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for caffeine in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for caffeine in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for omeprazole in the presence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
V/F for omeprazole in the absence of ecopipam | Up to Day 18
  Up to 38 blood samples will be collected at the indicated time points for pharmacokinetic analysis
Total concentration of bilirubin in the presence of ecopipam | Up to Day 13
  Bilirubin sampling will occur on Day 1 and Day 13
Total concentration of bilirubin in the absence of ecopipam | Up to Day 13
  Bilirubin sampling will occur on Day 1 and Day 13
Unconjugated concentration of bilirubin in the presence of ecopipam | Up to Day 13
  Bilirubin sampling will occur on Day 1 and Day 13
Unconjugated concentration of bilirubin in the absence of ecopipam | Up to Day 13
  Bilirubin sampling will occur on Day 1 and Day 13
Safety and tolerability as demonstrated by MOAA/S | Up to Day 55
  Safety and tolerability measures will be recorded at the indicated timepoints.
Safety and tolerability as demonstrated by C-SSRS | Up to Day 55
  Safety and tolerability measures will be recorded at the indicated timepoints.
Safety and tolerability as demonstrated by concomitant medications | Up to Day 55
  Safety and tolerability measures will be recorded at the indicated timepoints.
AEs with relatedness associated with dextromethorphan | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with IV midazolam | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with oral midazolam | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with dabigatran | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with pitavastatin | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with rosuvastatin | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with atorvastatin | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with bupropion | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with caffeine | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with omeprazole | Up to Day 55
  Subjects will be continually monitored for adverse events
AEs with relatedness associated with ecopipam | Up to Day 55
  Subjects will be continually monitored for adverse events
Absolute values of white blood cell (WBC) count (K/Ul) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of neutrophils, lymphocytes, monocytes, eosinophils, and basophils (10E3/uL) | Blood samples will be collected for the assessment of hematology parameters.
  Up to Day 25
Absolute values of platelets (K/uL) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of hematocrit (%) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of hemoglobin (g/dL) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of Red blood cell (RBC) count (M/uL) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Absolute values of blood sodium, magnesium, urea, phosphorus, potassium, and chloride (mg/dL) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of creatinine, calcium, glucose, and direct and total bilirubin (mg/dL) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of albumin and total protein (g/dL) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), and creatinine phosphokinase (CPK) (U/L) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Absolute values of urine specific gravity | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine pH | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine glucose | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine protein | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine blood | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine ketones | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine bilirubin, urobilinogen, and nitrite | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of urine leukocytes by dipstick | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in white blood cell (WBC) count (K/Ul) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in neutrophils, lymphocytes, monocytes, eosinophils, and basophils (10E3/uL) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in platelets (K/uL) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in hematocrit (%) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in hemoglobin (g/dL) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in Red blood cell (RBC) count (M/uL) | Up to Day 25
  Blood samples will be collected for the assessment of hematology parameters.
Change from Day -1 to Day of Discharge in blood sodium, magnesium, urea, phosphorus, potassium, and chloride (mg/dL) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in creatinine, calcium, glucose, and direct and total bilirubin (mg/dL) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in albumin and total protein (g/dL) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), and creatinine phosphokinase (CPK) (U/L) | Up to Day 25
  Blood samples will be collected for the assessment of clinical chemistry parameters.
Change from Day -1 to Day of Discharge in urine specific gravity | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine pH | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine glucose | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine protein | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine blood | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine ketones | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine bilirubin, urobilinogen, and nitrite (Milligrams per deciliter) | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Change from Day -1 to Day of Discharge in urine leukocytes by dipstick | Up to Day 25
  Urine samples will be collected for the assessment of urine parameters.
Absolute values of electrocardiogram (ECG) parameters: PR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) (Milliseconds) | Up to Day 25
  Twelve-lead ECGs will be obtained with the participant in a supine position after a rest of at least 5 minutes using an automated ECG machine. PR, QRS, QT, and QTcF intervals will be measured.
Change from pre-dose for the respective day in ECG parameters: PR, QRS, QT, and QTcF (Milliseconds) | Up to Day 25
  Twelve-lead ECGs will be obtained with the participant in a supine position after a rest of at least 5 minutes using an automated ECG machine. PR, QRS, QT, and QTcF intervals will be measured.
Absolute values of oral temperature (degrees Celsius) | Up to Day 25
  Temperature will be assessed as part of vital signs.
Change from pre-dose for the respective day in oral temperature (degrees Celsius) | Up to Day 25
  Temperature will be assessed as part of vital signs.
Absolute values of heart rate (beats/minute) | Up to Day 25
  Heart rate will be assessed as part of vital signs.
Change from pre-dose for the respective day in heart rate (beats/minute) | Up to Day 25
  Heart rate will be assessed as part of vital signs.
Absolute values of respiratory rate (breaths/minute) | Up to Day 25
  Respiratory rate will be assessed as part of vital signs.
Change from pre-dose for the respective day in respiratory rate (breaths/minute) | Up to Day 25
  Respiratory rate will be assessed as part of vital signs.
Absolute values of systolic blood pressure (SBP) and diastolic blood pressure (DBP) (mmHG) | Up to Day 25
  Blood pressure will be assessed as part of vital signs.
Change from pre-dose for the respective day in SBP and DBP (mmHG) | Up to Day 25
  Blood pressure will be assessed as part of vital signs.

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Clinical Research Services, LLC., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No